CLINICAL TRIAL: NCT04699058
Title: Sero-prevalence and Sero-conversion Study of Health Care Workers and Their Households, Democratic Republic of the Congo
Brief Title: COVID-19 Sero-prevalence Health Care Workers Kinshasa
Acronym: PRESTACOV
Status: Completed | Type: Observational
Sponsor: Institute of Tropical Medicine, Belgium (Other)
Collaborators: Institut National de Recherche Biomédicale. Kinshasa, République Démocratique du Congo (Other)
Responsible Party: Principal Investigator, Veerle Vanlerberghe, Principal Investigator, Institute of Tropical Medicine, Belgium
Other Study IDs: B3002020000144
Record Dates: First submitted 2020-12-04; First posted 2021-01-07 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-12

CONDITIONS: SARS-CoV Infection; Seroprevalence
MeSH Terms: conditions — Severe Acute Respiratory Syndrome

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — - For health care workers: Blood sample : a fingerprick , and one clotted blood tube to obtain serum (of 5 ml)
  - For Household members: Dried Blood spots: a fingerprick to collect minimum 3 - max 6 whole bloodspots
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Health care workers: questionnaire and COVID antibody test
  Interventions: Diagnostic Test: COVID-antibody test
- Household members: questionnaire and COVID antibody test
  Interventions: Diagnostic Test: COVID-antibody test

INTERVENTIONS:
Diagnostic Test: COVID-antibody test — Questionnaire and COVID-antibody test for all participants

SUMMARY:
This is a cohort study, in which the investigators will follow-up 650 health care workers (HCW) and a selection of their households (of COVID positive and COVID negative HCW) at baseline and in three follow-up surveys, with 4 to 6 weeks of time interval. The investigators will select HCW from different wards and different health care structures in 5 communes of Kinshasa. Additionally, in the first survey among HCW, the investigators will test with different diagnostic platform to evaluate the performance of serological tests in the African setting and the effect of malaria infection on the performance of tests.

An amendment is added to the protocol, stating an additional 2 surveys in april/June 2021 and October/November 2021 to evaluate impact of second wave and of vaccination campaign.

DETAILED DESCRIPTION:
Rationale:

There is no information on how intense transmission of COVID-19 happens in Kinshasa, partly due to a reduced laboratory capacity for polymerase chain reaction (PCR) confirmation of acute cases, and an aspecific presentation of clinical symptoms. The focus of this COVID-19 seroprevalence study on health care workers and their households, was based on the following rationale. Health care workers (HCW) are among the groups at higher risk as they are directly or indirectly exposed to COVID-19 patients. They also form a group of specific interest as they are in close contact to vulnerable patients at high risk for severe COVID-19. In addition, their illness or absence from work significantly affects the health system's ability to respond to the COVID-19 pandemic and retain its other essential functions. HCW are trained in infection prevention and control (IPC). However, it is likely that at least some of them will get infected either at their workplace(s) or elsewhere. In particular health facilities with limited access to personal protective equipment (PPE) and regular water and sanitation facilities, IPC could even potentially be hampered, resulting in an increased risk of infection transmission among HCW, from HCW to their patients as well as to their household members. Because of this crucial role played by HCW in the transmission chain, it is of utmost importance to assess the proportion of asymptomatic infections among them.

Aim of the study:

This study aims to investigate severe acute respiratory syndrome (SARS-CoV-2) seroprevalence and seroconversion among HCW in Democratic Republic of Congo (DRC) and their household members, including asymptomatic ones, in order to generate insights into the transmission dynamics as well as the clinical presentation of the disease.

Primary objectives

* Determine seroprevalence of SARS-CoV-2 infection among active HCW of hospitals and primary health care units of Kinshasa at T0;
* Determine seroprevalence of SARS-CoV-2 infection among household members of active HCW of hospitals and primary health care units of Kinshasa at T0;
* Determine incidence of SARS-CoV-2 seroconversions among HCW of hospitals and primary health care units of Kinshasa over a 3 months' time period;
* Determine SARS-CoV-2 seroconversion among household members of active HCW of hospitals and primary health care units of Kinshasa over a three months' time period.

Secondary objectives

* Identify work-related risk factors (infrastructural, availability of equipment and behavioral) for seroconversion of HCW;
* Identify socio-demographic and behavioral risk factors for seroconversion of household members;
* Determine the proportion of asymptomatic cases among seroconversions occurred during the study period among HCW as well as among their household members;
* Assess secondary attack rate among household members of symptomatic and asymptomatic HCW.
* To compare the performance of an in-house Luminex platform serologic diagnostic test, commercialized antibody ELISA test and an antibody rapid diagnostic test (RDT) against the gold standard serological test (neutralization) in tropical settings with intense cocirculation of malaria and other infectious diseases

Description: 650 HCW and 1000 household members will be surveyed at 4 time moments. At each moment, a questionnaire is filled exploring the professional and community risk exposure and the appearance of symptoms compatible with a COVID infection. At the same time, a serum sample is taken by the HCW and a 'dried blood spot' is done by the household members. These samples will be analyzed to verify if the participants were exposed to the SARS-CoV2 since the start of the epidemic. The use of a cohort will allow us to describe how the epidemic evolves over a 4 to 6 month period in Kinshasa, but will also make it possible to evaluate how the antibodies are waning or not waning over time.

An amendment is added to the protocol, stating an additional 2 surveys in april/June 2021 and October/November 2021 to evaluate impact of second wave and of vaccination campaign.

ELIGIBILITY:
Inclusion criteria:

For Both groups:

* Willing to provide written informed consent
* Being sick or having had COVID-19 is not an exclusion criterion

Health care workers

* Health care worker (all categories from specialist doctors to allied and auxiliary health workers) of the selected health services
* foreseen to be employed (or place of internship) for the next three months in he selected health facility

Household members

* Willing not to change the residence during the study period
* Household member of included Health care workers

Exclusion criteria: not giving consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Health care workers: All staff working in health care facilities of the selected health zones of Kinshasa: Lingwala, Bandalungwa, Limete, Ndjili and Lemba.
  Household members: All household members of participating Health care workers. Household members can be defined as the members of a household, which consists of a person or group of persons who live together in the same house, share the same housekeeping arrangements and usually eat meals together.
Sampling Method: Probability Sample
Enrollment: 1200 (Actual)
Dates: Start 2020-07-17 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
COVID antibody prevalence in Health care workers (serological test) | Month 2
  Antibody detection through ELISA and Luminex multiplex platform to estimate seroprevalence of SARS-CoV-2 infection among active HCW of hospitals and primary health care units of Kinshasa
COVID antibody prevalence in Household members (serological test) | Month 2
  Antibody detection through Luminex multiplex platform to estimate of SARS-CoV-2 infection among household members of active HCW of hospitals and primary health care units of Kinshasa
Seroconversion COVID Health care workers (serological test) | Month 6
  Serial antibody detection through Luminex multiplex platform to estimate incidence of SARS-CoV-2 seroconversions among HCW of hospitals and primary health care units of Kinshasa over a 5 months' time period
Seroconversion COVID household members (serological test) | Month 6
  Serial antibody detection through Luminex multiplex platform to estimate incidence of SARS-CoV-2 seroconversion among household members of active HCW of hospitals and primary health care units of Kinshasa over a five months' time period

SECONDARY OUTCOMES:
work-related exposure evaluated through a questionnaire and summarized as a score | Month 6
  the higher the score, the more exposed to the work-related risk factors (infrastructural, availability of equipment and behavioral); the higher the association is of a seroconversion with a higher score, the higher is the work-related exposure a risk factor for seroconversion.
behavioural risk factors (questionnaire), summarized as a score | Month 6
  the higher the score, the more exposed to risk behaviours (mobility, household); the higher the association is of a seroconversion with a higher score, the higher is the behaviour-related exposure a risk factor for seroconversion.

CONTACTS AND LOCATIONS:
Overall Officials: Veerle Vanlerberghe, PhD, Principal Investigator — ITG
Locations (1):
- Institut Nationale de recherche Biomédicale, Kinshasa, Democratic Republic of the Congo

IPD SHARING:
Plan to Share IPD: No
COVID-19 related information (sero-prevalence, individual status of infection, etc.) will not be made available openly to avoid stigmatisation, they will be made available upon request using a data sharing agreement to assure confidentiality for the individuals.